CLINICAL TRIAL: NCT01141179
Title: The Impact of Renal Impairment on the Pharmacokinetic and Pharmacodynamic of LEO 27847
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LEO 27847-S03
Record Dates: First submitted 2010-06-09; First posted 2010-06-10 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2013-11

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LEO 27847 (Experimental)
  Interventions: Drug: LEO 27847

INTERVENTIONS:
Drug: LEO 27847 — 2 mL (0.1 mg) dose of oral solution

SUMMARY:
The study will investigate the impact of reduced renal function on the pharmacokinetic and pharmacodynamic profile of LEO 27847. Volunteers with different degrees of renal impairment will be administered one dose of the investigational drug and then followed until investigational drug is eliminated from the body.

ELIGIBILITY:
Main Inclusion Criteria:

* Male and/or non-childbearing potential female, 18 years of age and older, healthy or with stable renal impairment (deemed stable by the referring physician for at least the last 4 weeks and not expected to change significantly during the next 3 months)
* BMI ≥18.0 and ≤ 42 kg/m2
* Patients with stable concomitant medical conditions
* Healthy subjects or patients with a creatinine clearance (at the time of screening) estimated using the formula of Cockcroft and Gault within the range of:

  * ≥ 50 to ≤ 80 mL/min (Mild Group: 8 subjects),
  * ≥ 30 to < 50 mL/min (Moderate Group: 8 subjects),
  * < 30 mL/min (Severe Group: 8 subjects).

Main Exclusion Criteria:

* Patients with renal transplants or currently on haemodialysis or peritoneal dialysis
* Clinically significant illness or surgery within 4 weeks prior to dosing
* Clinically significant ECG abnormalities or vital sign abnormalities at screening
* History of stroke, cerebrovascular disorder, coronary angioplasty and coronary bypass graft
* Clinically significant history or presence of any gastrointestinal pathology
* Use of medications other than their stable medications within 14 days prior to administration of investigational product or over-the-counter products within 7 days prior to administration of investigational product, except for:

  * multivitamins or vitamin D taken on a regular basis
  * topical products without systemic absorption
* Hemoglobin ≤ 90 g/L
* Serum total calcium (adjusted for albumin) level < 2.25 mmol/L
* Clinically significant history of congestive heart failure, cardiac dysfunction or liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-05; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
PK parameters | 1 week
  (AUC, Cmax)in each group of renal impairment

SECONDARY OUTCOMES:
PD parameters | 1 week
  (Calcium, phosphate, PTH), Vitamin D in each group of renal impairment

CONTACTS AND LOCATIONS:
Overall Officials: Richard Larouche, MD, Principal Investigator — Anapharm
Locations (1):
- Anapharm, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No